CLINICAL TRIAL: NCT04123327
Title: The Prevalence of Symptom Preoccupation and Its Role in AF-related Disability
Brief Title: Symptom Preoccupation in Atrial Fibrillation (AF) and Its Role in AF-related Disability
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Brjann Ljotsson, Associate Professor, Karolinska Institutet
Other Study IDs: Cross-sectional AF
Record Dates: First submitted 2019-10-09; First posted 2019-10-10 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2020-02

CONDITIONS: Atrial Fibrillation
Keywords: Symptom preoccupation; Atrial fibrillation; Quality of Life; Cardiac anxiety
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A cross-sectional study (N=400) will investigate the prevalence of symptom preoccupation and its role in AF-related disability. Subjectively-rated assessments will be gathered from 400 AF patients.

DETAILED DESCRIPTION:
In the present study we aim to investigate symptom preoccupation in patients with atrial fibrillation (AF) to further improve the understanding of the role of psychological factors in AF-related disability. A cross-sectional study (N=400) will investigate the prevalence of symptom preoccupation and its role in AF-related disability. Subjectively-rated assessments will be gathered from 400 AF patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Diagnoses with AF
* Able to read Swedish and access to computer

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients above 18 years of age and diagnosed with AF (paroxysmal, persistant or chronic)
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2019-12-24 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2020-10-10 (Actual)

PRIMARY OUTCOMES:
[Time Frame: From baseline to 12 weeks] Atrial Fibrillation Effect on Quality-of-Life (AFEQT) | Baseline
  AFEQT is an atrial fibrillation-specific measure that taps into the QoL-domains: symptoms, daily activities, treatment concern, and treatment satisfaction. The scale has 20 items, with the total score ranging from 0 (severe symptoms and disability) to 100 (no symptoms and disability), with responses provided on a seven-point rating scale from "no limitations/symptoms" to "severe limitations/symptoms".

SECONDARY OUTCOMES:
Cardiac Anxiety Questionnaire (CAQ) | Baseline
  It an 18-item scale that measures cardiac anxiety by three subscales fear (e.g., "When my heart is beating fast I get frightened" avoidance (e.g., I avoid exercise or other physical work) and attention (e.g., I pay attention to my heart beat). The responses are given on a four-point Likert scale ranging from 0 (never) to 4 (always), a greater score indicates greater cardiac anxiety.
Patient Health Questionnaire (PHQ-9) | Baseline
  Measures depressive symptoms on nine items scoring from 0 (not at all) to 3 (nearly every day) per item. Scores were categorized as follows: zero to minimal depressive symptoms (0-4), mild to moderate depressive symptoms (5-10), or severe depressive symptoms (10 or above).
The Generalized Anxiety Disorder (GAD-7) | Baseline
  The Generalized Anxiety Disorder (GAD-7) scale measures the severity of worry and anxiety. In healthy controls, the mean score was 4.9 (SD=4.8); a score of 10 or greater on the scale corresponds to a cut-off point for identifying cases of GAD.
Anxiety Sensitivity Index (ASI) | Baseline
  Measure of anxiety sensitivity
Bodily Sensation Questionnaire (BSQ) | Baseline
  Fear of bodily sensations
The University of Toronto Atrial Fibrillation Severity Scale (AFSS) | Baseline
  AFSS will assess AF symptoms and how affected the patient is by AF-specific symptoms such as dyspnea, palpitations etc. The AF symptom score ranges from 0-35 with a higher score indicating higher symptom severity.
The Symptoms Checklist, Frequency and Severity Scale (SCL) | Baseline
  SCL is a disease specific checklist used to measure AF-related symptoms (e.g., palpitations, dizziness) on two subscales: symptom severity (mild to extreme; 16 items, scores ranging from 0 to 48) and symptom frequency (never to always; 16 items, scores ranging from 0 to 64) over the past four weeks. Higher scores correlate with more frequent and severe symptoms.
Perceived Stress Scale (PSS-4) | Baseline
  To assess stress sensitivity and perception of stress. Each item is rated on a five-point scale and a higher score corresponds to more perceived stress.
World Health Organization Disability Assessment Schedule (WHODAS) | Baseline
  WHODAS is a reliable and well validated measure of general health and disability. We use the version consisting of 12-items evaluating six domains: cognition, mobility, self-care, getting along, life activities and life participation. Each item is rated on a 5-point scale, with higher scores indicating increased disability.
AF behaviors | Baseline
  Checklist of behaviors related to AF
Demographics | Baseline
  Demographics
Medical history | Baseline
  Comorbidities, medication, medical history

CONTACTS AND LOCATIONS:
Overall Officials: Brjánn Ljótsson, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Department of Clinical Neuroscience, Karolinska Institutet, Stockholm, Sweden